CLINICAL TRIAL: NCT05675813
Title: Guidance-04：T-cell Lymphoma Series：A Genotype-guided Therapy in Newly Diagnosed Patients With Peripheral T-cell Lymphoma （THEORY Study）
Brief Title: Genotype-guided Treatment in Newly Diagnosed PTCL
Acronym: THEORY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); Peking University Third Hospital (Other); Wuhan TongJi Hospital (Other); West China Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Anhui Provincial Cancer Hospital (Other); The First Affiliated Hospital of Soochow University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Beijing Tongren Hospital (Other); Peking University People's Hospital (Other); Sun Yat-sen University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhao Weili, Vice President, Ruijin Hospital, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Guidance-04 (NHL-016)
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Biomarker-driven; Genetic subtypes; Complete response rate; Phase 1/2; Precision medicine
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T1: CHOP+selinexor+5-Azacitidine (CHOPX2) vs CHOP (Experimental): Phase I: Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the first cycle. If tumor NGS indicates T1 genetic subtype, for the remaining 5 cycles, they will receive 5-Azacitidine ih d-7-d-1 and selinexor 40mg or 60mg qw (d-7, 1, 8) by traditional "3+3" dose escalation methods and decide RP2D of selinexor.
  Phase II: Patients will receive CHOP for the first cycle. If tumor NGS indicates T1 genetic subtype, then 1:1 randomized to experimental (CHOPX2) or standard CHOP regimen for 5 cycles of every 21-day cycle.
  Interventions: Drug: CHOP+selinexor+5-Azacitidine; Drug: standard CHOP
- T2: CHOP+duvelisib+5-Azacitidine vs CHOP (Experimental): Phase I: Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the first cycle. If tumor NGS indicates T2 genetic subtype, for the remaining 5 cycles, they will receive 5-Azacitidine ih d-7-d-1 and duvelisib 25mg or 50mg bid (d1-14) by traditional "3+3" dose escalation methods and decide RP2D of duvelisib.
  Phase II: Patients will receive CHOP for the first cycle. If tumor NGS indicates T1 genetic subtype, then 1:1 randomized to experimental (CHOPX2) or standard CHOP regimen for 5 cycles of every 21-day cycle.
  Interventions: Drug: CHOP+duvelisib+5-Azacitidine; Drug: standard CHOP
- T3: CHOP+chidamide+tislelizumab （CHOPX2）vs CHOP (Experimental): Phase I: Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the first cycle. If tumor NGS indicates T3 genetic subtype, for the remaining 5 cycles, they will receive tislelizumab 200mg d0 ivgtt and chidamide 20mg or 30mg biw (d1,4,8,11) by traditional "3+3" dose escalation methods and decide RP2D of chidamide.
  Phase II: Patients will receive CHOP for the first cycle. If tumor NGS indicates T3 genetic subtype, then 1:1 randomized to experimental (CHOPX2) or standard CHOP regimen for 5 cycles of every 21-day cycle.
  Interventions: Drug: CHOP+chidamide+tislelizumab; Drug: standard CHOP

INTERVENTIONS:
Drug: CHOP+selinexor+5-Azacitidine — Phase I: Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the first cycle. If tumor NGS indicates T1 genetic subtype, for the remaining 5 cycles, they will receive 5-Azacitidine ih d-7-d-1 and selinexor 40mg or 60mg qw (d-7, 1, 8) by traditional "3+3" dose escalation methods and decide RP2D of selinexor.
  Phase II: Patients will receive CHOP for the first cycle. If tumor NGS indicates T1 genetic subtype, then 1:1 randomized to experimental (CHOPX2) or standard CHOP regimen for 5 cycles of every 21-day cycle.
  Arms: T1: CHOP+selinexor+5-Azacitidine (CHOPX2) vs CHOP
Drug: CHOP+duvelisib+5-Azacitidine — Phase I: Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the first cycle. If tumor NGS indicates T2 genetic subtype, for the remaining 5 cycles, they will receive 5-Azacitidine ih d-7-d-1 and duvelisib 25mg or 50mg bid (d1-14) by traditional "3+3" dose escalation methods and decide RP2D of duvelisib.
  Phase II: Patients will receive CHOP for the first cycle. If tumor NGS indicates T1 genetic subtype, then 1:1 randomized to experimental (CHOPX2) or standard CHOP regimen for 5 cycles of every 21-day cycle.
  Arms: T2: CHOP+duvelisib+5-Azacitidine vs CHOP
Drug: CHOP+chidamide+tislelizumab — Phase I: Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the first cycle. If tumor NGS indicates T3 genetic subtype, for the remaining 5 cycles, they will receive tislelizumab 200mg d0 ivgtt and chidamide 20mg or 30mg biw (d1,4,8,11) by traditional "3+3" dose escalation methods and decide RP2D of chidamide.
  Phase II: Patients will receive CHOP for the first cycle. If tumor NGS indicates T3 genetic subtype, then 1:1 randomized to experimental (CHOPX2) or standard CHOP regimen for 5 cycles of every 21-day cycle.
  Arms: T3: CHOP+chidamide+tislelizumab （CHOPX2）vs CHOP
Drug: standard CHOP — Patients in this arm will receive cyclophosphamide 750 mg/m² IV, doxorubicin 50 mg/m² IV, and vincristine 1.4 mg/m² IV (maximum 2 mg) on day 1, and prednisone 100 mg/day PO on days 1-5 of every 21-day cycle for the 6 cycles.

SUMMARY:
This study includes Phase I and Phase II stages. Phase I is an open-label trial to confirm RP2D of oral targeted agents in three genetic subtypes. Phase II is a multicenter, prospective, randomized, open-label, controlled trial to evaluate the efficacy and safety of genotype-guided targeted agents plus cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP-X2) versus cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) in patients with peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL) is a heterogeneous disease with dismal outcomes. Standard CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisolone) chemotherapy is still the most widely used front-line treatment of PTCL except Brentuximab-CHP application in anaplastic large cell lymphoma (ALCL). The CR rate ranges from 31%-56% in different studies with different PTCL histology compositions. With the exception for ALCL-anaplastic lymphoma kinase (ALK)-positive, the 5-year overall survival (OS) rate is approximately 30%-40% for most subtypes of PTCL patients in current situation, remaining as the unmet medical needs in this disease. Based on genetic subtypes in PTCL, and our previous study exploring targeted agents plus CHOP based on genetic mutations (Guidance-03 study), we conducted this multicenter, prospective, randomized, open-label, controlled trial to evaluate the efficacy and safety of genotype-guided targeted agents plus CHOP (CHOP-X2) versus cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) in patients with PTCL. It includes phase I and phase II stages. Patients will receceived stardard CHOP for the first cycle and then obtain the genetic subtypes from tumor NGS befor Cycle 2. In phase I, recommended phase 2 dose (RP2D) of oral targeted agents will be confirmed by traditional "3+3" dose escalation methods. In phase II, patients will receive standard CHOP for the first cycle and then 1:1 be randomized to CHOPX2 or CHOP regimen in each genetic subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed Peripheral T-cell lymphoma
* Availability of archival or freshly collected tumor tissue before study enrollment enough for NGS
* Evaluable lesion by PET-CT or CT scan
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life expectancy greater than or equal to (>/=) 3 months
* Informed consent

Exclusion Criteria:

* Patients with ALCL and cutaneous TCL
* Patients with central nervous system (CNS) lymphoma
* History of malignancies except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrolled cardio- and cerebro-vascular disease, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
* Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

Neutrophils<1.0×10^9/L Platelets<75×10^9/L (Platelets<50×10^9/L in case of bone marrow involvement) ALT or AST is 2.5 times higher than the upper limits of normal (ULN), AKP and bilirubin are 1.5 times higher than the ULN.

Creatinine is 1.5 times higher than the ULN.

* HIV-infected patients
* Active hepatitis infection
* Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
* Pregnant or lactation
* Other medical conditions determined by the researchers that may affect the study For T3 should exclude patiens with active autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) for Phase I | DLT time window (28 days from Cycle 2)
  Recommended Phase 2 Dose (RP2D) for Phase I of oral targeted agents in each genetic subtypes by traditional "3+3" dose escalation methods
Complete response rate (CRR) for Phase II | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days])
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 4 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China